CLINICAL TRIAL: NCT01343732
Title: Tolerability, Safety and Efficacy of the HAC-Coil Deep Transcranial Magnetic Stimulation in Medication Resistance Obsessive Compulsive Disorder (OCD) Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OCD-DTMS-1
Record Dates: First submitted 2011-04-11; First posted 2011-04-28 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-01

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

ARMS (4):
- healthy volunteeres (No Intervention): this arm will undergo only EEG measurement
- real - low frequency (Active Comparator): this arm will receive DTMS treatment with low frequency
  Interventions: Device: Deep TMS
- real - high frequency (Active Comparator): this arm will receive DTMS treatment with high frequency
  Interventions: Device: Deep TMS
- sham - low / high frequency (Sham Comparator): this arm will receive DTMS sham treatment with low or high frequency
  Interventions: Device: Deep TMS

INTERVENTIONS:
Device: Deep TMS — deep transcranial magnetic stimulation
  Arms: real - high frequency; real - low frequency; sham - low / high frequency

SUMMARY:
The purpose of this study is to test whether the combination of deep transcranial magnetic stimulation (DTMS) treatment with customary medication for obsessive compulsive disorder (OCD) patients is effective than treatment that include only medication.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. Men and Women 18-65 years of age.
3. Diagnosed as suffering from OCD according to DSM-IV.
4. Patients having OCD of at least moderate severity (YBOCS score of 20 or above).
5. Patients are maintained on an medication at steady dosages for at least 8 weeks before study entry and for the duration of the trail.
6. Negative answers on safety screening questionnaire for transcranial magnetic stimulation.
7. According to the treating physician the patients is compliant with taking medication.
8. Capable and willing to provide informed consent.
9. Able to adhere to treatment schedule.
10. Patients that participate in behavioral therapy, will be in the maintaining stage and not in the active or intensive stage.

Exclusion Criteria:

1. Any other Axis I diagnosis as the primary diagnosis.
2. History of epilepsy or seizure (EXCEPT those therapeutically induced by ECT) or history of such in first degree relatives).
3. OCD patients that have only symptoms of hoarders)
4. patients with Suicidal tendencies, or the patients is diagnosed as having a Suicidal tendencies by the treating physician.
5. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
6. History of head injury necessitating cranial surgery or prolonged coma.
7. History of any metal in the head including the eyes and ears (outside the mouth).
8. Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
9. History of frequent or severe headaches.
10. History of migraine.
11. History of significant hearing loss.
12. Individuals with a significant neurological disorder or insult including, but not limited to:

    Any condition likely to be associated with increased intracranial pressure Space occupying brain lesion History of cerebrovascular accident Transient ischemic attack within two years Cerebral aneurysm Dementia Parkinson's disease Huntington's chorea Multiple sclerosis
13. History of substance abuse including alcoholism within the past 6 months (except nicotine and caffeine).
14. Inadequate communication with the patient.
15. Participation currently in another clinical study or enrolled in another clinical study within 30 days prior to this study.
16. Participants who suffer from an unstable physical, systemic and metabolic disorders such as instabilized blood pressure or acute, unstable cardiac disease.
17. Women who are breast-feeding.
18. Known or suspected pregnancy.
19. Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Y-BOCS Scale (Yale-Brown Obsessive Compulsive Disorder) | the primary outcome will be measure at day, 8, 22, 31, and 33

CONTACTS AND LOCATIONS:
Overall Officials: Yossef Zohar, Prof., Principal Investigator — Sheba Medical Center, ramat-gan, Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Carmi L, Alyagon U, Barnea-Ygael N, Zohar J, Dar R, Zangen A. Clinical and electrophysiological outcomes of deep TMS over the medial prefrontal and anterior cingulate cortices in OCD patients. Brain Stimul. 2018 Jan-Feb;11(1):158-165. doi: 10.1016/j.brs.2017.09.004. Epub 2017 Sep 6. PMID 28927961